CLINICAL TRIAL: NCT06693297
Title: Immediate Versus Conventional Loading of Early Placed Dental Implant Supporting Single Crowns: a Randomized Controlled Trial
Brief Title: Immediate Versus Conventional Loading of Early Placed Dental Implant Supporting Single Crowns
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jordan (Other)
Collaborators: Straumann Group (Unknown); MegaGen (Unknown)
Responsible Party: Principal Investigator, Mohammad AL-Rababáh, Associate Professor, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10/2024/22294
Record Dates: First submitted 2024-11-03; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Dental Implant
Keywords: dental implant; thread design; immediate loading; conventional loading; early placement

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional loading of early placed implants (Active Comparator): Early placed implants ( within 16 weeks of healing after Extraction of a tooth) will be conventionally loaded ( at least 8 weeks after implant placement )
  Interventions: Device: Immediate loading of early placed implants; Device: Conventional loading of early placed implants
- Immediate loading of early placed implants (Experimental): Early placed implants (within 16 weeks of tooth extraction) will be loaded immediately with provisional screw retained crown
  Interventions: Device: Immediate loading of early placed implants; Device: Conventional loading of early placed implants

INTERVENTIONS:
Device: Immediate loading of early placed implants — Implants with active thread design will be used. The implants placed will be randomly allocated into either immediate loading or conventional loading group.
Device: Conventional loading of early placed implants — Definitive loading of early placed implants upon successful osteointegration (after 8 weks)

SUMMARY:
This study focuses on examining the efficacy and clinical performance of immediate loading of early placed single implants.

The aim of the randomized controlled trial is to compare between two loading protocols (immediate versus conventional) of early placed implants (Type 2-3A) in terms of clinical, radiographic, and patient-reported outcomes.

Null hypothesis: There will be no significant differences in implant survival/success, stability, radiographic marginal bone level, and patient reported outcomes between immediately or conventionally loaded and early placed implants.

DETAILED DESCRIPTION:
Study design:

This study is designed as a parallel group randomized controlled trial with an allocation ratio of 1:1.

The (PICO) study design: population will be patients from Jordan University Hospital aged 18 years or older, requiring single tooth replacement (molar or premolar) with dental implants, with sufficient bone volume and controlled oral hygiene. The intervention group will receive immediate loading of early placed implants (within 1 week), while the comparator group will receive conventional loading (after more than 8 weeks). The primary outcome is changes in marginal bone levels, and the secondary outcomes include implant primary osseointegration, stability, patient satisfaction, and various complications.

Both groups will receive early placed implants after 8-12 weeks of healing (Type 2-3A placement). The surgical procedure will follow standardized protocols, with no variations between groups other than the loading time.

Blinded assessors will perform radiographic and clinical evaluations at designated follow-up visits: at implant placement, definitive loading, 6 months, and 1 year. Ethical approval is obtained prior to study commencement, and all participants will provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18 years or older
2. requiring single tooth replacement with dental implants in presence of four bone walls (mandible or maxilla)
3. having adequate bone volume
4. controlled oral hygiene
5. having agreed to take part in the study and willing to comply with the study protocol and follow-up visits

Exclusion Criteria:

1. Any systemic condition that might jeopardize implant surgery
2. history of radiation therapy to the head and neck region
3. history of bisphosphonate therapy or other medications that may affect bone metabolism
4. smoking more than 10 cigarettes/day
5. history of bruxism or parafunctional habits
6. localized/generalized periodontitis
7. patients in need of bone grafting
8. any known allergy or hypersensitivity to implant materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Marginal bone level changes | Baseline (day of implant placement), at definitive loading (more than 8 weeks post-placement for the conventional loading group, within 1 week post-placement for the immediate loading group), and at 1-year follow-up post-loading.
  Marginal bone level changes by standardized periapical radiographs.

SECONDARY OUTCOMES:
Implant failure rate | 1 year
  defined as implant removal
Implant stability | Baseline (day of implant placement), at definitive loading (more than 8 weeks post-placement for the conventional loading group, within 1 week post-placement for the immediate loading group)
  Osstell readings
Midfacial mucosal level | at time of delivery of definitive prosthesis (more than 8 weeks post-placement for the conventional loading group, within 1 week post-placement for the immediate loading group) and one-year follow-up
  as measured by periodontal probe
Pink and white esthetic scores | at time of delivery of definitive prosthesis (more than 8 weeks post-placement for the conventional loading group, within 1 week post-placement for the immediate loading group) and one-year follow-up
Patient Satisfaction | after 6 months and 1 year of placements
  To be assesses by oral health impact profile-14 (OHIP-14), The scale includes 14 items covering various aspects of oral health-related quality of life, Score Range: from 0 to 56, Higher OHIP-14 scores indicate a worse outcome, representing a greater negative impact of oral health issues on quality of life, while lower scores suggest a better outcome or less impact on the individual's daily life.
Biological, estehtic and technical complications | 1 year
  (infection, implant mobility, or prosthesis-related issues) assessed by expert prosthodontist who is blind to the nature of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Jordan University Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No